CLINICAL TRIAL: NCT06813794
Title: The Effect of Message Framing in Diabetic Foot Self-Management on Diabetic Foot Care Behaviors and Self-Efficacy: a Randomized Controlled Trial
Brief Title: The Effect of Message Framing in Diabetic Foot Self-Management
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mehtap KAVURMACI, Prof., Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B.30.2.ATA.0.01.00/327
Record Dates: First submitted 2025-01-13; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus
Keywords: message framing; Diabetic foot care; Self-efficacy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Gain-Framed) (Experimental): Participants receive gain-framed messages emphasizing the benefits of proper foot care.
  Interventions: Behavioral: Gain- Framed Messages
- Control Group (No Intervention): Participants will receive neutral messages about diabetic foot care.
- Group 2 (Loss-Framed) (Experimental): Participants receive loss-framed messages highlighting the risks of inadequate foot care.
  Interventions: Behavioral: Lost Framed Messages

INTERVENTIONS:
Behavioral: Gain- Framed Messages — Patients will be recruited to whatsapp group based on gain framing about diabetic foot care skills. Gain framing messages and videos will be delivered to patients via whatsapp 3 times a week for 3 months.
  Arms: Group 1 (Gain-Framed)
Behavioral: Lost Framed Messages — Patients will be included in whatsapp group based on Lost framing about diabetic foot care skills. Patients will receive loss framing messages and videos 3 times a week for 3 months via whatsapp.
  Arms: Group 2 (Loss-Framed)

SUMMARY:
This study aims to assess how effective gain- and loss-framed messages are in improving diabetic foot care behaviors and increasing self-efficacy levels compared to routine foot care messages.

Study Design:

A randomized controlled trial with three groups:

Experimental Group 1 (Gain-Framed): Participants receive gain-framed messages emphasizing the benefits of proper foot care.

Experimental Group 2 (Loss-Framed): Participants receive loss-framed messages highlighting the risks of inadequate foot care.

Control Group (Routine Messaging): Participants receive standard foot care messages without specific framing.

Participants:

Diabetic patients recruited from Experimental Group 1, Experimental Group, and Control Group 3. Inclusion criteria include adults diagnosed with diabetes who are at risk for diabetic foot complications.

Intervention:

Over a period of three months, participants will receive WhatsApp messages three times a week.

Gain-Framed Messages: Emphasize positive outcomes, such as preventing foot ulcers by wearing appropriate footwear.

Loss-Framed Messages: Highlight negative consequences, such as the increased risk of foot infections from improper foot care.

Messages will include supportive images and videos to enhance engagement and understanding.

Outcome Measures:

Primary Outcomes:

Foot Care Behavior: Assessed using The Foot Care Behavior Scale. Self-Efficacy: Measured by the Diabetic Foot Care Self-Efficacy Scale Secondary Outcomes: Comparative effectiveness between gain-framed and loss-framed messages.Long-term behavioral changes post-intervention.

Significance:

This study seeks to determine the most effective messaging strategy to promote diabetic foot care, potentially informing future interventions to reduce the incidence of diabetic foot complications.

DETAILED DESCRIPTION:
Title: The Effect of Message Framing on Self-Efficacy and Foot Care Behaviors in Diabetic Foot Care: A Randomized Controlled Study

Abstract:

This study aims to examine the effect of message framing on self-efficacy and foot care behaviors in diabetic foot care. Evaluating the impact of message framing on self-efficacy and foot care behaviors is crucial in reducing the economic burden of diabetic foot on healthcare services while simultaneously improving patients' quality of life and daily functionality. The results of this study are expected to contribute to interventions aimed at enhancing self-efficacy in diabetic foot care and preventing diabetic foot complications.

Study Setting and Population:

Patients will be recruited through diabetes-related social media groups. Eligible participants who agree to participate will be contacted via WhatsApp, where they will receive framed messages.

Study Design and Methodology:

This study is designed as a three-arm randomized controlled trial.

Population and Sample: The study population consists of patients following diabetes-related social media groups. The sample will include individuals meeting the inclusion criteria and consenting to participate between May 15, 2024, and May 15, 2025. Participants will be randomly assigned to one of three groups: Experimental Group 1, Experimental Group 2, and Control Group 3. A three-month intervention will be implemented.

Sample Size Calculation: The sample size was determined using the G*Power 3.1.9.6 program. A three-group, two-measurement (pretest, posttest) design was considered. Based on an effect size of 0.50, a significance level of α = 0.05, and a power of 1-β = 0.80, the required sample size for each group was calculated as 49. Considering possible data loss, the sample size was increased by 10%, resulting in 54 participants per group and a total of 162 participants.

Randomization: Simple random sampling (lottery method) will be used. The lottery draw will be conducted by an independent person with no contact with the participants.

Intervention Procedure:

Participants in all groups will receive an online questionnaire via Google Forms, including a Patient Information Form, the Diabetic Foot Self-Efficacy Scale, and the Foot Care Behavior Scale.

Experimental Group 1: Participants will receive gain-framed messages about diabetic foot care via a WhatsApp group. Three times a week for three months, they will be sent gain-framed messages and videos. For example, a message emphasizing proper footwear and socks will state: "Wearing appropriate shoes and socks that reduce foot friction helps prevent foot ulcers caused by vascular damage." Healthy foot images and videos will accompany the messages.

Experimental Group 2: Participants will receive loss-framed messages via WhatsApp. Three times a week for three months, they will receive loss-framed messages and videos. An example message will be: "Wearing inappropriate shoes and socks that increase foot friction may lead to poor foot care and a higher risk of foot ulcers." Images of infected feet and videos of patients receiving treatment for diabetic foot complications will be shared.

Control Group 3: Participants will receive neutral messages regarding foot care without specific message framing. For example, they will receive the message: "You should wear appropriate shoes and socks to prevent foot friction."

At the end of the intervention, the Diabetic Foot Self-Efficacy Scale and Foot Care Behavior Scale will be re-administered.

Data Collection Tools:

Patient Information Form: Collects demographic data (age, gender, education level, date of diabetes diagnosis, presence of foot complications).

Diabetic Foot Self-Efficacy Scale: Developed by Bonnie Elliott Quarles in 2005 to assess diabetic patients' perceived ability to perform foot care activities. The Turkish validity and reliability study was conducted by Biçer and Enç in 2011. The 9-item scale is scored on a visual scale from 0 (not confident) to 10 (very confident), with a total score range of 0-90. A higher score indicates higher self-efficacy (Cronbach's α = 0.86).

Foot Care Behavior Scale: Originally developed by Borges in 2007 as the Foot Care Observation Guide and later adapted by Biçer and Enç in 2011. This 15-item Likert-type scale measures foot care behaviors, ranging from 1 (never) to 5 (always). The total score ranges from 15 to 75, with higher scores indicating better foot care behaviors (Cronbach's α = 0.83).

Limitations:

The study is limited to information measured by the surveys and to patients with internet access who voluntarily participate.

Ethical Considerations:

Ethical approval will be obtained from the Ethics Committee of Atatürk University Faculty of Medicine. Institutional permissions will be sought from relevant hospitals. Written informed consent will be obtained from participants.

Data Collection and Storage:

Data will be collected through Google Forms via WhatsApp after obtaining informed consent from voluntary participants.

Data Analysis:

Survey responses will be analyzed using SPSS software. Statistical analyses will include comparisons of pretest and posttest scores across groups using appropriate statistical methods.

Conclusion:

This study aims to evaluate the effectiveness of message framing on diabetic foot care self-efficacy and behaviors. Findings are expected to contribute to the development of targeted interventions that enhance diabetic foot care practices, reduce healthcare costs, and improve patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 55 years.
* Individuals diagnosed with diabetes for at least six months.
* Individuals without diabetic foot ulcers or amputations.
* Individuals without any communication disorders or psychiatric illnesses.
* Individuals who are members of a social media platform.
* Individuals who can use a smartphone and have internet access.
* Individuals willing to participate in the study.
* Individuals with at least a primary school education.

Exclusion Criteria:

* Individuals diagnosed with diabetes (This criterion seems unclear; please clarify if it should refer to a specific diabetes-related condition).
* Individuals with diabetic foot ulcers or amputations.
* Individuals with any communication disorders or psychiatric illnesses.
* Individuals without access to a smartphone or the internet.
* Individuals with malingering disorders.
* Individuals who are illiterate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Diabetic Foot Care Self-Sufficiency Level | 3 months
  Diabetic Foot Care Self-Efficacy Scale will be applied to the patients in Experimental Group 1, Experimental Group 2 and Control Group 3.
  Primary Outcome: Change in Diabetic Foot Care Self-Efficacy Score from baseline to 3 months.
  Measurement Timepoints: Baseline (Pretest) and 3-Month Follow-up (Posttest).The lowest score that can be obtained from the Diabetic Foot Care Self-Efficacy Scale is 0 and the highest score is 90. As the score obtained from the scale increases, the level of diabetic foot self-efficacy increases.
Assessment of Foot Care Behavior | 3 month
  Foot Care Behavior Scale will be applied to the patients in Experimental Group 1, Experimental Group 2 and Control Group 3. Primary Outcome: Change in Foot Care Behavior Scale from baseline to 3 months.
  Measurement Timepoints: Baseline (Pretest) and 3-Month Follow-up (Posttest).The lowest score of the Foot Care Behavior scale is 15 and the highest score is 75. The increase in the scale score indicates that the individual's self-care behaviors are better

CONTACTS AND LOCATIONS:
Overall Officials: Mehtap Kavurmacı, Prof, Study Director — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gao R, Guo H, Liu Y, Pang Y, Zhang X, Lian X, Yu T, Zhu L, Li F. The effects of message framing on self-management behavior among people with type 2 diabetes: A randomized controlled trial. Int J Nurs Stud. 2023 Jun;142:104491. doi: 10.1016/j.ijnurstu.2023.104491. Epub 2023 Mar 17. PMID 37059032
- See also: The International Working Group on the Diabetic Foot: Stories and Numbers Behind Three Decades of Evidence-Based Guidelines for the Management of Diabetes-Related Foot Disease — https://pmc.ncbi.nlm.nih.gov/articles/PMC10786793/